CLINICAL TRIAL: NCT02730195
Title: Combination of Pioglitazone and Tyrosine Kinase Inhibitor (TKI) in Relapsed Chronic Myeloid Leukemia Following a First TKI Discontinuation
Brief Title: Pioglitazone and Tyrosine Kinase Inhibitor in Treating Patients With Relapsed Chronic Myeloid Leukemia
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, William Blum, Principal Investigator, Emory University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00086670; NCI-2016-00248 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); Winship3121-15 (Other: Emory University/Winship Cancer Institute)
Record Dates: First submitted 2016-03-29; First posted 2016-04-06 (Estimated); Results first posted 2019-01-09 (Actual); Last update posted 2019-01-09 (Actual); Status verified 2018-12

CONDITIONS: Chronic Myelogenous Leukemia, BCR-ABL1 Positive; Recurrent Chronic Myelogenous Leukemia, BCR-ABL1 Positive
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive | interventions — Pioglitazone; Tyrosine Kinase Inhibitors

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Pioglitazone & TKI therapy (Experimental): Patients receive pioglitazone PO QD on days 1-28. Patients also start or continue the same tyrosine kinase inhibitor (TKI) therapy at the pre-discontinuation doses. Courses repeat every 28 days for 6 months in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Pioglitazone; Drug: Tyrosine Kinase Inhibitor (TKI)

INTERVENTIONS:
Drug: Pioglitazone — Given PO
  Other Names: Actos; Pioglitazone Hydrochloride
Drug: Tyrosine Kinase Inhibitor (TKI) — Given TKI therapy
  Other Names: Protein Tyrosine Kinase Inhibitors; PTK Inhibitors; TK Inhibitors

SUMMARY:
This phase II trial studies how well pioglitazone hydrochloride and tyrosine kinase inhibitor (TKI) therapy works in treating patients with chronic myeloid leukemia (CML) that has come back after a period of improvement (relapsed) after a first TKI discontinuation. TKI may stop the growth of cancer cells by blocking certain enzymes need for cell growth. Although TKI therapies are effective against CML, there are residual cancer cells called leukemia stem cells that are able to hide from TKIs. Pioglitazone is a drug approved by the Food and Drug Administration to treat diabetes and has been shown in laboratory studies to increase CML stem cell death when given together with TKI therapy. Giving pioglitazone with TKI therapy may be effective in treating patients with CML.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess safety of the combination of pioglitazone (PIO) and TKI in CML subjects who experience a loss of major molecular response (MMR) following a first TKI discontinuation.

II. To assess survival without loss of MMR following a second TKI discontinuation in subjects who achieve or maintain < molecular response (MR)^4.5 with the combination PIO and TKI administered for at least 6 months.

OUTLINE:

Patients receive pioglitazone orally (PO) once daily (QD) on days 1-28. Patients also start or continue the same TKI therapy at the pre-discontinuation doses. Courses repeat every 28 days for 6 months in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every month for 3 months, every 3 months for 1 year, and then every 6 months for 4 years.

ELIGIBILITY:
Inclusion Criteria:

* Chronic myeloid leukemia (CML) in any phase
* Philadelphia chromosome positive acute lymphoblastic leukemia
* Loss of major molecular response (MMR) following a first TKI discontinuation trial
* Serum bilirubin < 1.5 x upper limit of normal values
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) < 2.5 x upper limit of normal values
* Females of child bearing potential must agree to abstain from sexual activity or to use a medically approved contraceptive measure/regimen during and for 3 months after the treatment period; women of child bearing potential must have a negative urine pregnancy test at the time of enrollment; acceptable methods of birth control include oral contraceptive, intrauterine device, transdermal/implanted or injected contraceptives and abstinence
* Males must agree to abstain from sexual activity or agree to utilize a medically-approved contraception method during and for 3 months after the treatment period
* Patient requiring anti-diabetic medications to manage hyperglycemia are eligible. Adjustments of other anti-diabetic agents will be made with close monitoring of blood glucose
* Informed consent
* Be able and willing to comply with study visits and procedures

Exclusion Criteria:

* Known loss of complete cytogenetic response (CCyR) by marrow cytogenetic or blood fluorescence in situ hybridization (FISH) for breakpoint cluster region (BCR)- v-abl Abelson murine leukemia viral oncogene homolog 1 (ABL1)
* Loss of complete hematologic response (CHR)
* Participation in another clinical trial with any investigative drug within 30 days prior to study enrollment
* Chronic graft-versus-host disease requiring systemic immunosuppression post-allogeneic hematopoietic stem cell transplantation
* Cardiovascular disease: history of congestive heart failure, myocardial infarction in the 6 months preceding study entry, symptomatic cardiac arrhythmia requiring treatment
* History of bladder cancer
* Gross (visible) hematuria
* Known history of osteoporosis
* Known history of macular edema
* Known history of ABL1-domain mutation that predicts resistance to the discontinued TKI
* Significant medical or psychiatric disorder that would interfere with consent, study participation, or follow-up
* Known allergy to pioglitazone
* Pregnant or breastfeeding
* Use of thiazolidinedione (TZD) within 28 days prior to enrollment
* Significant gastrointestinal condition that could potentially impair the absorption or disposition of the drug
* Uncontrolled peripheral edema (2+ or more) of any etiology
* Active cancer that requires therapy in the form of chemotherapy or radiation

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2016-05; Primary Completion 2018-07 (Actual); Study Completion 2018-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William Blum, MD, Principal Investigator — Emory University
Locations (1):
- Emory University/Winship Cancer Institute, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Groups:
- Pioglitazone & TKI Therapy: Patients receive pioglitazone PO once a day (QD) on days 1-28. Patients also start or continue the same tyrosine kinase inhibitor (TKI) therapy at the pre-discontinuation doses. Courses repeat every 28 days for 6 months in the absence of disease progression or unacceptable toxicity.
  Pioglitazone: Given PO
  Tyrosine Kinase Inhibitor (TKI): Given TKI therapy
Period: Overall Study
Arm/Group | Pioglitazone & TKI Therapy
Started | 9
Completed | 8
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Pioglitazone & TKI Therapy
Number analyzed (Participants) | 9
Age, Customized [Count of Participants; unit: Participants]
  30-39 years old | 1
  40-49 years old | 2
  50-59 years old | 1
  60-69 years old | 4
  70-79 years old | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 9
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 6
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 9

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Adverse Events (AEs), Graded According to Common Terminology Criteria for Adverse Events Version 4.03
Description: The AE incidence will be described. An AE is any untoward medical occurrence in a subject or clinical investigation subject administered a pharmaceutical product which does not necessarily have to have a causal relationship with this treatment. AEs will be assessed through scheduled assessments and subject reported diaries.
Time Frame: Up to 30 days after the end of treatment
Measure: Number; unit: events
Arm/Group | Pioglitazone & TKI Therapy
Number analyzed (Participants) | 9
events
  Number of Grade 1 Events | 41
  Number of Grade 2 Events | 0
  Number of Grade 3 Events | 0
  Number of Grade 4 Events | 0
  Number of Grade 5 Events | 0

2. Primary Outcome: Proportion of Subjects Who Achieve and Maintain Major Molecular Response (MMR) Following a Second Discontinuation of TKI Using Blood Quantitative Reverse Transcription Polymerase Chain Reaction (qRT-PCR) for Breakpoint Cluster Region-Abelson1 (BCR-ABL1)
Description: The proportion of subjects that has reappearance of BCR-ABL1 will be described. Descriptive statistics that will summarize the changes in BCR-ABL1 testing over time will be presented. Subgroup analyses will be performed by baseline potential prognostic factors. Subgroups will include: age, gender, race, underlying diagnosis, and other disease-related prognostic factors (disease status).
Time Frame: Up to 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Pioglitazone & TKI Therapy
Number analyzed (Participants) | 9
Participants | 8

3. Secondary Outcome: Proportion of Subjects Who Lose MMR Following Discontinuation of Pioglitazone and TKI Using Blood qRT-PCR for BCR-ABL1
Description: The proportion of subjects that has reappearance of BCR-ABL1 will be described. Descriptive statistics that will summarize the changes in BCR-ABL1 testing over time will be presented. Loss of MMR is defined as a BCR-ABL1 > 0.1% by qRT-PCR confirmed within a week and associated with a rise in the titer on a confirmatory test obtained 4 weeks later (European Leukemia Net definition). Subgroup analyses will be performed by baseline potential prognostic factors. Subgroups will include: age, gender, race, underlying diagnosis, and other disease-related prognostic factors (disease status).
Time Frame: Up to 3 years
Measure: Count of Participants; unit: Participants
Arm/Group | Pioglitazone & TKI Therapy
Number analyzed (Participants) | 9
Participants | 7

ADVERSE EVENTS:
Time Frame: Up to 30 days after the end of treatment
Arm/Group | Pioglitazone & TKI Therapy
All-Cause Mortality (participants affected / at risk) | 0/9
Serious Adverse Events (participants affected / at risk) | 0/9
Other Adverse Events (participants affected / at risk) | 7/9
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pioglitazone & TKI Therapy (N=9)
Edema limbs (General disorders) | 5
Fatigue (General disorders) | 2
Edema face (General disorders) | 1
Night sweats (General disorders) | 1
Diarrhea (Gastrointestinal disorders) | 2
Nausea (Gastrointestinal disorders) | 2
Constipation (Gastrointestinal disorders) | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 1
Muscle cramps (Musculoskeletal and connective tissue disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1
Headache (Nervous system disorders) | 1
Paresthesia (Nervous system disorders) | 1
Peripheral sensory neuropathy (Nervous system disorders) | 1
Urinary frequency (Renal and urinary disorders) | 3
Urine discoloration (Renal and urinary disorders) | 1
Creatinine increased (Investigations) | 1
Platelet count decreased (Investigations) | 1
White blood cell decreased (Investigations) | 1
Irregular menstruation (Reproductive system and breast disorders) | 1
Nipple tenderness (Reproductive system and breast disorders) | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1
Upper respiratory infection (Respiratory, thoracic and mediastinal disorders) | 1
Alopecia (Skin and subcutaneous tissue disorders) | 1
Bruising (Skin and subcutaneous tissue disorders) | 1
Anemia (Blood and lymphatic system disorders) | 1
Palpitations (Cardiac disorders) | 1
Vertigo (Ear and labyrinth disorders) | 1

LIMITATIONS AND CAVEATS:
Study was terminated early due to previous principal investigator leaving institution.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-04-05): https://cdn.clinicaltrials.gov/large-docs/95/NCT02730195/Prot_SAP_000.pdf